CLINICAL TRIAL: NCT05306405
Title: Comparative Study Between Using Only Vaginal Misoprostol and Using Vaginal Misoprostol and Estradiol Cream for Induction of Labour
Brief Title: Comparative Study Between Only Vaginal Misoprostol and Vaginal Misoprostol and Estradiol Cream
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Maher, Resident of Obstetrics and Gynecology at Al-Delengat General Hospital, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2022-02-18; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Cervix; Pregnancy
Keywords: cervical dilatation, Uneffaced cervix, closed os
MeSH Terms: interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vaginal misoprostol (Active Comparator): only vaginal misoprostol 25 μg tablets will be applied for induction of laour
  Interventions: Drug: Vaginal Tablet
- combined vaginal misoprostol and estradiol (Active Comparator): vaginal misoprostol 25 μg (Vagiprost) tablets with vaginal estradiol 150 ml cream will be applied for induction of laour
  Interventions: Drug: Vaginal Tablet

INTERVENTIONS:
Drug: Vaginal Tablet — Misoprostol alone will be repeated every 4 h in both groups for a maximum of 5 doses, reaching Bishop score >8, rupture of membranes or occurrence of labor pain.
  Cervical evaluation will be done using Bishop's score. A score < 5 will be taken as unfavorable Cervix will be termed as ripped when Bishop's score equal 8 or more.
  The endpoint of the study will be initiation of active phase of 1st stage of labor which commence from 6cm to full cervical dilatation
  Other Names: vaginal misoprostol and vaginal estradiol

SUMMARY:
To compare the safety and effectiveness of vaginal misoprostol with combined vaginal misoprostol and estradiol for induction of labour in unfavorable cervix

DETAILED DESCRIPTION:
Induction of labour (IOL) is the process of initiating contractions of pregnant persons who are currently not in labour, to help them achieve vaginal delivery within 24 to 48 hours. Cervical ripening is one of the methods that used for labour induction; it is "the use of pharmacological or other means to soften, efface, or dilate the cervix to increase the likelihood of a vaginal delivery". The two major techniques for cervical ripening are mechanical interventions (e.g. insertion of balloon catheters), and application of pharmacological agents (e.g. prostaglandins). Prostaglandins are one of the preferred methods for cervical ripening, including the agents dinoprostone and misoprostol

. By the mid of-1980s prostaglandins had become established as the most effective pharmacological agents for inducing labour when the cervix is unripped. The vaginal route was found to be the most acceptable, providing good efficacy and acceptability for the parturient and it is the preferred choice now.

During the past 15 years the introduction of misoprostol, the prostaglandinsE1(PGE1) which, unlike prostglandinsE2 (PGE2), is stable at room temperature and it is effective if it was taken orally, has been the major focus of attention for labour induction. It is also considerably cheaper than the alternative prostaglandin.

With the ever-increasing concentrations of estrogen in the maternal circulation leading to term pregnancy, the belief that this could be a trigger for the onset of spontaneous labour led the studies to explore estrogens for the induction of labour.

Estradiol gel gives extra--amniotic, endocervical or vaginally or estradiol intramuscularly and estradiol gel extra-amniotic have been shown to produce some improved cervical favorability with minimal myometrial stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age36:41 weeks.
* Singleton pregnancy.
* Absence of labour pain.
* Living fetus with cephalic presentation.
* Fetal weight < 4 k.gs.
* No previous uterine surgical procedures.
* No liquor abnormalities.
* Bishop score < 5.

Exclusion Criteria:

* - Multiple gestations. one of the contraindications of induction of labor as it may cause rupture of the uterus.
* Liquor abnormalities.one of contraindications of induction of labor as it may cause fetal distress.
* Abnormal umbilical artery Doppler indices or non-stress test as these indicate fetal distress.
* Fetal weight > 4 kgs.as macrosomia is an indication of caesarean section for fear of shoulder dystocia .
* Previous uterine surgery.contraindication of labor induction for fear of rupture uterus.
* Asthmatic patient or women with allergy to prostaglandins or steroidal.
* Non-vertex presentation.contraindication of labor induction as it may cause rupture uterus.
* Fetal or maternal complications that might cause cesarean section.
* Intrauterine fetal death.often induction of labor in women with a dead fetus is performed before term when the uterus may be less responsive to uterotonics than it is at term and this will affect the results of the study

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Induction of labour with closed cervix | from 0 hours to 14 hours after induction of labour
  assessment of uterine contractions and cervical opening of the pregnant females who are currently not in labour, to help them to reach normal vaginal delivery process.

SECONDARY OUTCOMES:
The Whole Delivery time after induction of labour. | from 0 hours to the end of the delivery
  The whole time from induction to the end of vaginal labour with complications that may arise as:
  -uterine hyperstimulation, postpartum hemorrhage, rupture of the uterus and neonatal morbidity, fetal distress, and fetal hypoxia.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No